CLINICAL TRIAL: NCT05247385
Title: Platelet Aggregation and Adenosine Levels Among Patients With Stable Chronic Coronary Artery Disease Taking Ticagrelor or Prasugrel
Brief Title: Platelet Aggregation and Adenosine Levels Among Patients Taking Ticagrelor or Prasugrel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jose Carlos Nicolau, Director Coronary Care Unit, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4086/14/066
Record Dates: First submitted 2022-01-04; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prasugrel group (Active Comparator): Prasugrel (60mg loading dose, followed by 10 mg QD for 15 days)
  + Ticagrelor placebo (Placebo loading dose followed by two pills a day)
  Interventions: Drug: Prasugrel; Drug: Ticagrelor
- Ticagrelor group (Active Comparator): Ticagrelor (180mg loading dose, followed by 90 mg BID)
  + Prasugrel placebo (Placebo loading dose followed by one pill a day)
  Interventions: Drug: Prasugrel; Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Compared platelet inhibition and adenosine levels at baseline and after 15 days
Drug: Ticagrelor — Compared platelet inhibition and adenosine levels at baseline and after 15 days

SUMMARY:
Prospective, single-center, double blind, double dummy, randomized trial. Platelet function tests and adenosine levels were assessed at baseline and 15 days after taking Ticagrelor with Prasugrel placebo or Prasugrel with Ticagrelor placebo in stable patients with coronary artery disease

DETAILED DESCRIPTION:
This was a prospective, double blinded, randomized trial that compared platelet inhibition and adenosine levels with ticagrelor (180mg loading dose, followed by 90 mg BID) versus prasugrel (60mg loading dose, followed by 10 mg QD) .

Patients were eligible if they were between 18 and 75 years old, were on aspirin without P2Y12 inhibitor at baseline and > 1 year after documented ACS. Platelet aggregation was compared with the Multiplate ADP® assay, performed at baseline and after 15 days on study medication. Adenosine plasma levels were measured with high performance liquid chromatography at the same time points

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 75 years old
* were on aspirin
* without P2Y12 inhibitor at baseline
* > 1 year after documented acute coronary syndrome

Exclusion Criteria:

* use of oral anticoagulation or P2Y12 at baseline
* Weight < 60kg
* History of tia or stroke
* Any coagulation disorders
* Refuse to sign the written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
To compare platelet inhibition between the two groups (ticagrelor and prasugrel) | 15 days
  Platelet aggregation was compared with the Multiplate ADP® assay at baseline and after 15 days on study medication
To compare adenosine levels between the two groups (ticagrelor and prasugrel) | 15 days
  Adenosine plasma levels were measured at baseline and after 15 days with high performance liquid chromatography at the same time points

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor) / University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No